CLINICAL TRIAL: NCT06928571
Title: A Hybrid Effectiveness/ Implementation Trial Using Online Tools to Increase Weight Loss Among Primary Care Patients
Brief Title: Using Online Tools to Increase Weight Loss in Primary Care
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202400390; R01DK137092 (NIH)
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: Statistician/analyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect4Health Engage (Experimental): Receive Connect4Health Engage
  Interventions: Behavioral: Connect4Health Engage
- Connect4Health Discover (Active Comparator): Receive Connect4Health Discover
  Interventions: Behavioral: Connect4Health Discover

INTERVENTIONS:
Behavioral: Connect4Health Engage — Intervention focused on motivating and guiding patients to use empirically supported, freely available online tools for weight loss.
  Arms: Connect4Health Engage
Behavioral: Connect4Health Discover — Educational control - information about healthy eating and physical activity
  Arms: Connect4Health Discover

SUMMARY:
The goal of the proposed project is to test the effectiveness of an intervention (Connect4Health Engage) focused on motivating and guiding patients to use empirically supported, freely available online tools for weight loss. A randomized trial will be conducted in primary care clinics. Fifteen to twenty PCPs will be recruited, followed by 453 patients. Patients will complete either the 52-week Connect4Health Engage intervention or Connect4Health Discover, an educational control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* BMI ≥ 30 kg/m2 based on self-report body weight and height, OR BMI 27-29.9 kg/m2 with a weight related comorbidity of hypertension, type 2 diabetes, pre-diabetes, dyslipidemia, or obstructive sleep apnea, gastroesophageal reflux disease, or coronary artery disease.
* Self-report weight ≤ 375 lbs (the maximum weight that BodyTrace scales can accurately detect is 397 lbs, thus 375 lbs provides a buffer to allow detection of at least 20 lbs weight gain).
* Has valid email address in EHR
* Has an appointment scheduled with enrolled PCP about 30-45 days after IDR query
* Speaks and reads English
* Has either WiFi internet access at home or a phone or tablet with a data plan.

Exclusion Criteria:

* BMI≥ 45 kg/m2.
* Currently enrolled in structured weight loss treatment
* In past month, has been actively participating in a weight loss focused online community (i.e., posting or reading content).
* Currently tracking food intake 3 days per week
* Pregnant or planning to become pregnant in the next 6 months
* Currently breastfeeding (or pumping breastmilk) 3 times per day or more.
* Currently undergoing treatment for cancer or has active cancer
* Had cardiovascular event in the past 60 days
* Inpatient psychiatric treatment in the past 6 months
* Eating disorder in past 5 years
* Congestive heart failure resulting in recent (past 6 months) hospitalization or contributing to difficulty breathing or difficulty doing daily activities.
* Dementia diagnosis
* Bariatric surgery in the past year or currently undergoing evaluation for bariatric surgery
* Type 1 Diabetes
* Currently taking prescription medication for weight loss
* Inability to stand on body weight scale independently
* Impaired hearing
* Unable to read content on websites without assistance
* Planning to move out of the region in the next 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Proportion achieving ≥ 3% weight loss | 52 weeks
  Proportion of patients achieving ≥3% weight loss

SECONDARY OUTCOMES:
Weight stability at 78 weeks | 78 weeks
  Proportion of individuals who do not exceed 3% weight gain from baseline.
Weight change at 52 weeks (continuous) | 52 weeks
  Weight change from baseline to week 52 in kgs (continuous)
Weight change at 78 weeks (continuous) | 78 week
  Weight change from baseline to week 78 in kgs (continuous)
Weight stability at 52 weeks | 52 weeks
  Proportion of individuals who do not exceed 3% weight gain from baseline at 52 weeks.
Minutes of moderate-to-vigorous physical activity per week at 52 weeks | 52 week
  Minutes of moderate-to-vigorous physical activity per week as measured using the International Physical Activity Questionnaire (IPAQ) (continuous measure MET minutes per week)
Minutes of moderate-to-vigorous physical activity per week at 78 weeks | 78 weeks
  Description: Minutes of moderate-to-vigorous physical activity per week as measured using the International Physical Activity Questionnaire (IPAQ) (continuous measure MET minutes per week)
Servings per day of fruits and vegetables (52 weeks) | 52 weeks
  Number of servings per day of fruits and vegetables measured by Eating at America's Table Study (EATS) fruit and vegetable screener.
Servings per day of fruits and vegetables (78 weeks) | 78 weeks
  Number of servings per day of fruits and vegetables measured by Eating at America's Table Study (EATS) fruit and vegetable screener.
Percentage of energy from fat (52 weeks) | 52 weeks
  Percent of energy from fat measured using NCI Percentage Energy from Fat Screener measure
Percentage of energy from fat (78 weeks) | 78 weeks
  Percent of energy from fat measured using NCI Percentage Energy from Fat Screener measure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data will be shared with other researchers. Researchers will need to complete a Data Use Agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available within six months of completing data collection, or at the time of the first associated publication, whichever comes first.
Access Criteria: The data and documentation will only be made available to users under a Data Use Agreement (DUA) that ensures commitments to using the data only for research purposes; to protecting identification of any individual subject; to securing the data using appropriate computer technology; and to destroying or returning the data to us after analyses are completed. To protect the privacy and confidentiality of participants and to ensure appropriate use of these data, the deidentified data will be shared in a restricted repository to be made available to qualified researchers who submit an application and execute a DUA with the appropriate participant protections. Consistent with our institution's IRB requirements, data will be available for up to five years following the study's completion.